CLINICAL TRIAL: NCT02056106
Title: Task Shifting Model of Depression Treatment to Unleash HIV Public Health Benefits
Brief Title: Comparative Trial of Antidepressant Treatment Models in HIV Care in Uganda
Acronym: INDEPTH-Uganda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Glenn Wagner, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH098996 (NIH)
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Depression
Keywords: depression, Uganda, HIV, task-shifting, condom use, adherence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical acumen (Active Comparator): Depression diagnosis and antidepressant treatment provided based on clinical acumen of primary care providers trained to provide depression care.
  Interventions: Drug: antidepressant therapy
- Protocolized Arm (Active Comparator): Structured, algorithm-based protocol that guides depression diagnosis and antidepressant treatment
  Interventions: Drug: antidepressant therapy

INTERVENTIONS:
Drug: antidepressant therapy

SUMMARY:
This study compares two models for implementing antidepressant treatment in 10 HIV clinics in Uganda. Using a cluster randomization, 5 clinics implement a task-shifting, protocolized model, and 5 others rely on clinical acumen. The protocolized model includes (1) routine depression screening at each clinic visit for all adult patients by trained expert patients at triage, (2) training nurses to diagnose depression and prescribe and monitor antidepressant treatment using an algorithm-based protocol, and (3) monthly supervision and monitoring by hired study psychiatrists. The clinical acumen model also includes routine depression screening and ongoing supervision, but it relies on the clinical acumen of trained primary care providers to further evaluate and treat patients who show signs of depression at screening, as opposed to a structured protocol. The primary aim is to test the hypothesis that the nurse-driven protocolized model will result in greater uptake of antidepressant treatment and better quality of depression care outcomes. The study will also test the hypotheses that treatment of depression results in improved HIV treatment adherence, work functioning and consistent condom use.

DETAILED DESCRIPTION:
The study evaluates a task-shifting approach to depression treatment that uses an algorithm-based, nurse-driven model for managing antidepressant treatment in 10 Ugandan HIV clinics. The model will include (1) case identification facilitated by routine depression screening at each clinic visit for all patients, (2) training nurses to assist primary care providers in implementing antidepressant treatment by performing the initial evaluation, monitoring symptoms and side effects, and making algorithm-based dose recommendations, and (3) layers of supervision and monitoring by psychiatric specialists to ensure safety and quality of care. This model will be implemented at 5 randomly selected clinics (protocolized arm), while 5 other clinics will be selected to also use routine depression screening but will rely on primary care providers to decide whether to further evaluate and treat depression (clinical acumen arm). At each site, random samples of 150 patients (total n=1500) who have screened positive for possible depression will be followed for 12 months. We will compare the two arms on depression evaluation, uptake of antidepressant treatment, and change in depression (treatment response). We will also examine the relationship between change in depression and key economic and public health outcomes (e.g. work status, condom use, HIV treatment adherence).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* screens positive for depression (scores > 2 on PHQ-2)
* medically stable
* client at the HIV clinic (and hence, HIV positive)

Exclusion Criteria:

* active acute opportunistic infection
* about to start HIV antiretroviral therapy or started antiretroviral therapy within past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Depression diagnostic evaluation | baseline, Month 6, Month 12
  Whether or not the Patient Health Questionnaire (PHQ-9) was administered to assess severity of depression
Antidepressant prescription | baseline, Month 6, Month 12
  Whether or not antidepressants were prescribed; this variable will be analyzed among the subset of patients categorized as depressed based on PHQ-9 > 9
Depressive symptoms | past 2 weeks at Month 6 and Month 12
  depressive symptoms present at Month 6 and Month 12 (in comparison to baseline) to assess treatment response; PHQ-9 will be used to measure depressive symptoms

SECONDARY OUTCOMES:
Consistent condom use | past 6 months prior to baseline, Month 6, Month 12
  A single likert scale item will be used to assess condom use in the past month; a single item will also be used to assess whether condom was used during last event of sexual intercourse
ART adherence | past month prior to baseline, Month 6 and Month 12
  single variable to rate adherence to ART over the past month on scale of 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, PhD, Principal Investigator — RAND
Locations (1):
- health care facilities receiving technical assistance from Mildmay Uganda, Wakiso, Mpigi, Luwero, Mityana Districts, Uganda

REFERENCES:
- [Derived] Wagner GJ, Ngo V, Goutam P, Glick P, Musisi S, Akena D. A Structured Protocol Model of Depression Care versus Clinical Acumen: A Cluster Randomized Trial of the Effects on Depression Screening, Diagnostic Evaluation, and Treatment Uptake in Ugandan HIV Clinics. PLoS One. 2016 May 11;11(5):e0153132. doi: 10.1371/journal.pone.0153132. eCollection 2016. PMID 27167852
- [Derived] Wagner GJ, Ngo V, Glick P, Obuku EA, Musisi S, Akena D. INtegration of DEPression Treatment into HIV Care in Uganda (INDEPTH-Uganda): study protocol for a randomized controlled trial. Trials. 2014 Jun 25;15:248. doi: 10.1186/1745-6215-15-248. PMID 24962086